CLINICAL TRIAL: NCT01031433
Title: Assessment of Craving in Nicotine-Dependent Patients With Schizophrenia Using Virtual Reality
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909449; 09-DA-N449
Record Dates: First submitted 2009-12-11; First posted 2009-12-14 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2012-07-18

CONDITIONS: Nicotine Dependence
Keywords: Tobacco Craving; Virtual Reality; Schizophrenia; Smoking
MeSH Terms: conditions — Tobacco Use Disorder; Schizophrenia; Smoking

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* The prevalence of cigarette smoking among individuals with schizophrenia is noticeably higher than in the general population, and smoking cessation attempts frequently are unsuccessful in this population. Little is known about the effects of cigarette/nicotine craving in individuals with schizophrenia. Researchers are interested in learning more about how craving affects people with schizophrenia and developing new ways to treat cravings and improve the effectiveness of smoking cessation therapies and treatments.
* In recent years, virtual reality (VR) has been studied to determine whether it can be used to induce craving by using life-like cue settings. VR cues involving cigarette use, including images of cigarettes and scent cues of tobacco smoke, may be used to elicit craving in smokers. Researchers are interested in learning more about how individuals with schizophrenia respond to specific VR cues and settings.

Objectives:

* To determine the feasibility of using a contextual real-world paradigm using virtual reality involving cigarette smoking in people with schizophrenia.
* To examine if virtual reality cues will elicit craving in smokers with schizophrenia.

Eligibility:

- Current smokers (five or more cigarettes per day for at least 1 year) between 18 and 45 years of age who have been diagnosed with schizophrenia/schizoaffective disorder.

Design:

* The study will involve three sessions, with an initial screening visit, a test session, and a follow-up session.
* Screening visit: Participants will be screened with a medical and psychiatric history, and will answer questions about smoking history, current smoking habits and craving patterns, and general anxiety levels. This session will also introduce participants to the operation and use of the VR equipment. Participants who are comfortable using the VR system will return within 2 days for the test session.
* Test session: Participants will use the VR equipment to view neutral scenes and scenes that are designed to elicit cravings for cigarettes. After viewing each scene, participants will answer questions about their overall mood, anxiety levels, and any cigarette cravings they may have.
* Follow-up session: Participants will return 1 week after the VR session to answer questions about mood, anxiety levels, and current smoking habits and craving patterns.

DETAILED DESCRIPTION:
Objective:

Nicotine use is high in people with schizophrenia; however, interventions to aid in smoking cessation have not been overwhelmingly successful. Craving, particularly situational craving, is one reason people relapse. Craving paradigms in people with schizophrenia need to be optimized in order to test new treatments on craving measures in this population. Thus, the purpose of this study is to determine the feasibility and effects of virtual reality cues on craving intensity for smoking in patients with schizophrenia

Study population:

We will enroll 25 smokers with a DSM IV diagnosis of schizophrenia with the goal of obtaining a total of 16 completers.

Design:

This study uses a comparison-controlled, within-subject design. All subjects will undergo a baseline assessment and acclimation period and then participate in an experimental condition in which four cues will be presented in separate rooms in the VR program. These include two smoking cues and two neutral cues in four different rooms. A follow up session for craving and symptom assessments will occur one week after the experimental session.

Outcome Measures:

During the Cue trials the Cigarette Craving Visual Analogue Scale (CCVAS), a four-item scale, and the Tobacco Craving Questionnaire-Short Form (TCQ-SF)will be administered to measure cigarette craving during the virtual reality session. At the end of each of the 4 cues (neutral, smoking cue with no interaction, smoking cue with interaction, neutral) participants will be asked about craving. The CCVAS will be projected into the VR environment and participants will respond via hand controller. To assess mood status, the Mood form will also be administered at baseline as well as at the end of each of the 4 cues. Before and after the experimental session participants will also be rated on the Brief Psychiatric Rating Scale (BPRS), Schedule for the Assessment of Negative Symptoms (SANS), side effects, and the State-Trait Anxiety Inventory (STAI). The Immersion Questionnaire and Imagery Realism Presence Questionnaire (PQ) will be given at the conclusion of the experimental session. During the experiment participants will be monitored for physiological reactivity (heart rate, blood pressure, and skin conductance response) to cues of smoking as well as neutral cues measured. Additionally, subjects will be assessed before and after the experimental session

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. 18-55 year old males and females
  2. Currently smokes at least 5 cigarettes per day
  3. Current DSM-IV diagnosis of schizophrenia and stable medication regimen
  4. Medically healthy as determined by screening criteria
  5. Urine cotinine level greater than or equal to 100 ng/ml (NicAlert reading greater than or equal to 3)
  6. Agrees to wear a head mounted display (HMD) for up to 45 minutes
  7. Participant able to complete the Evaluation to Sign Consent (ESC) with minimum score of 80 percent on ESC.

EXCLUSION CRITERIA:

1. Interest in reducing or quitting tobacco use within the past 3 months
2. Treatment for tobacco dependence in the past 3 months
3. Use of nicotine replacement products, bupropion, or varenicline in the past 3 months as an aid to quit or reduce smoking.
4. DSM-IV diagnosis of active alcohol or substance abuse in the past 1 month or dependence within the past 6 months
5. Current use of serotonin reuptake inhibitors or any medication that would interfere with the protocol in the opinion of MAI
6. History of head injury, seizures, or stroke
7. Pregnant, nursing, or planning to become pregnant during the study
8. Positive urine toxicology screen for substances other than those used for therapeutic purposes: participants who have an initial positive urine toxicology screen for substances other than those used for therapeutic purposes will have the opportunity to return within two weeks for a second toxicology screen. If at that time the results are again positive, the participants will be excluded.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2009-07-28; Study Completion 2012-07-18

PRIMARY OUTCOMES:
During the Cue trials the Cigarette Craving Visual Analogue Scale (CCVAS) will be administered to measure cigarette craving during the virtual reality session.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Heishman, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- University of Maryland at Baltimore/MPRC, Catonsville, Maryland, United States

REFERENCES:
- [Background] Andreasen NC. Negative symptoms in schizophrenia. Definition and reliability. Arch Gen Psychiatry. 1982 Jul;39(7):784-8. doi: 10.1001/archpsyc.1982.04290070020005. PMID 7165477
- [Background] Bordnick PS, Graap KM, Copp H, Brooks J, Ferrer M, Logue B. Utilizing virtual reality to standardize nicotine craving research: a pilot study. Addict Behav. 2004 Dec;29(9):1889-94. doi: 10.1016/j.addbeh.2004.06.008. PMID 15530734
- [Background] Carter BL, Tiffany ST. Meta-analysis of cue-reactivity in addiction research. Addiction. 1999 Mar;94(3):327-40. PMID 10605857